CLINICAL TRIAL: NCT06833970
Title: Investigation of Color Changes in the Teeth of Individuals Using Different Toothpastes During Orthodontic Treatment
Brief Title: Toothpastes With Different Contents and Tooth Color
Status: Completed | Type: Observational
Sponsor: Taner OZTURK, DDS, MS (Other)
Responsible Party: Sponsor-Investigator, Taner OZTURK, DDS, MS, Associate Professor, TC Erciyes University
Organization: TC Erciyes University (Other)
Other Study IDs: 2024/253
Record Dates: First submitted 2025-01-09; First posted 2025-02-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: White Spot Lesion of Tooth; Tooth Color; Dentistry; Orthodontic Appliances, Fixed
Keywords: Tooth color change; Toothpaste; Dentifrice

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1 Control: Individuals using a toothpaste (Colgate) with a fluoride content of 1450 ppm, which is frequently reported in the literature and used commercially internationally, will be included. Whether the patients continue to use the relevant toothpaste will be confirmed with information provided by the patient at each session of orthodontic treatment.
  Interventions: Other: Colgate use; Device: Fixed orthodontic treatment
- Group 2 Lactoperoxidase: Individuals using a toothpaste (Curaprox) with lactoperoxidase and content of 1450 ppm fluoride, which is frequently reported in the literature and used commercially internationally, will be included. Whether the patients continue to use the relevant toothpaste will be confirmed with information provided by the patient at each session of orthodontic treatment.
  Interventions: Other: Curaprox use; Device: Fixed orthodontic treatment
- Group 3 Non-fluoridate: Individuals using a biocompatible mineral and natural enzyme toothpaste (ROCS) instead of the fluoride, sodium lauryl sulphate and paraben content reported in the literature and commercially used internationally will be included. Whether the patients continue to use the relevant toothpaste will be verified with the information provided by the patient at each session of orthodontic treatment.
  Interventions: Other: ROCS use; Device: Fixed orthodontic treatment

INTERVENTIONS:
Other: Colgate use — An evaluation of Colgate total toothpaste currently in use will be provided.
  Groups: Group 1 Control
Other: Curaprox use — An evaluation of Curaprox toothpaste currently in use will be provided.
  Groups: Group 2 Lactoperoxidase
Other: ROCS use — An evaluation of ROCS toothpaste currently in use will be provided.
  Groups: Group 3 Non-fluoridate
Device: Fixed orthodontic treatment — For standard fixed orthodontic treatment, orthodontic brackets and mechanics will be applied.

SUMMARY:
This study aims to investigate the color tone and fluorescence changes that may occur during fixed orthodontic treatment with brackets in patients' teeth using toothpaste with different properties. The study will include routinely taken three-dimensional models, fluorescence photographs, gingival index, periodontal index, ICDAS II, and DMFT index records of patients who have received orthodontic treatment at Erciyes University Faculty of Dentistry and who have been using the same toothpaste for a long time. Three different toothpaste groups were determined to be included in the study. These toothpastes will be examined in three groups: those with fluoride effect, those containing lactoperoxidase, and those without fluoride, which are routinely used by patients. It was decided that there would be 15 individuals in each group in case individuals were excluded from the clinical study to be conducted. As a result, 45 patients, 15 in each group, will be included in the study. This study will use digital models obtained by scanning the upper and lower jaws of the patients included using an intraoral scanner (3shape TRIOS). The reason for this is to evaluate whether there will be a change in the color of the patient's teeth during the orthodontic treatment process by comparing them with the records taken in the later stages of the treatment. Photographic records of the patients will also be taken with the Quantitative Laser-Induced Fluorescence (QLF) device. With this device, the fluorescence color change that occurs on the tooth surfaces will be examined.

DETAILED DESCRIPTION:
Background

Studies examining the effectiveness of toothpastes on white spot lesions seen with fluorescence color change during orthodontic treatment are available in the literature in vitro and in vivo. Since in vivo studies are still insufficient in number, some records showing oral hygiene and periodontal health were added to the records to be taken from patients in this study. Literature studies have taken similar records, such as an in-vivo study by Hoffman et al., which evaluated the effects of two different toothpastes on white spot lesions and included plaque index and gingival index records taken from patients in 3-month periods. Another study by Kirschneck et al. investigated the effectiveness of fluoride pastes and varnishes on white spot lesions and recorded ICDAS index and gingival index values from patients at 4, 12, and 20 weeks after the beginning of treatment. Karabekiroğlu et al. compared a group using only fluoride toothpaste with a test group in which 10% casein phosphopeptide-amorphous calcium phosphate (CPP-ACP) paste was applied topically, including records such as ICDAS 2, DMFT and DMFS index, and QLF records. In the study to be conducted, comprehensive records such as DMFT index, gingival index, plaque index, ICDAS 2 index, QLF records, and color analysis of the teeth obtained from digital models taken with the intraoral scanning device will be collected from patients at specified periods. Since the tooth color tones determined with the 3Shape Trios device, the intraoral scanning device used in the clinic, are based on the Vita scale, a reference article in the literature will be used to facilitate statistical analysis. The images of the scanning records will be transferred to Adobe Photoshop, and the color values will be converted to L.a.b. and ∆E parameters. This conversion allows for the numerical equivalent of the color tones, making statistical analysis easier. The demineralization values of 10 teeth, excluding the molars in the upper jaw, will be measured using the QLF device's own software.

Methods

The study will include routinely taken three-dimensional models, fluorescence photographs, gingival index, periodontal index, ICDAS II, and DMFT index records of patients who have received orthodontic treatment at Erciyes University Faculty of Dentistry and who have been using the same toothpaste for a long time.

Three different toothpaste groups to be included in the study were determined. These toothpastes will be examined in three groups as those routinely used by patients with fluoride effect, those containing lactoperoxidase, and those without fluoride. The number of patients in the groups was determined using the G*Power (Ver. 3.1.9.7, Heinrich Heine University, Dusseldorf, Germany) power analysis program, based on DF values of the control group followed up with standard toothpaste in a study by Bröchner et al. in 2011. According to the two-way student t-test power analysis with d=1.384 effect value, 95% power, and alpha=0.05 parameters, at least 12 individuals should be in each group. To account for possible exclusions from the clinical study, 15 individuals were included in each group. As a result, a total of 45 patients, with 15 patients in each group, will be included in the study. The patients will be randomly assigned to three groups using a free randomization program mentioned in the literature. The purpose of this method is to ensure that the distribution of the patients into groups is random. Traditionally, dental models, intraoral and extraoral photographs, radiographic images, and clinical measurement records will be taken from patients before orthodontic treatment. Digital models obtained by scanning the upper and lower jaws using an intraoral scanner (3shape TRIOS) will be used. The purpose of this is to evaluate whether there will be a change in tooth color during the orthodontic treatment process by comparing them with records taken in the later stages of treatment. Photographic records will also be taken with a Quantitative Laser-Induced Fluorescence (QLF) device, which will be used to examine fluorescence color changes on the tooth surfaces. Patients who have started their treatment after the records are taken will be divided into three groups, and each group will use the assigned toothpaste throughout the treatment. The group using only fluoride-containing toothpaste will serve as the control group. The study will evaluate upper incisors, canines, first, and second premolars. Periodontal and gingival index measurements will be taken as part of the routine examination before, during, and at the end of orthodontic treatment. ICDAS II and DMFT tooth decay presence scoring methods will be performed through intraoral examination during photo record collection.

Statistical Evaluation

Statistical evaluations will be performed with the R-based JAMOVI analysis program. Statistical comparisons of changes in the number of white spot lesions on teeth evaluated over time will be made using analysis of variance (ANOVA) for repeated measurements within each group. Suppose a statistically significant difference is observed between measurement times within each group. In that case, paired samples t-tests will be used to determine at which time points the difference is statistically significant. Whether a statistically significant difference exists between groups, between times, and in the group-time interaction will be evaluated separately using multiple analyses of variance (ANOVA). If a statistically significant difference is observed between groups or time points, Tukey HSD multiple comparison tests will be used to identify the specific differences. The statistical significance value will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients in permanent dentition,
* No tooth extractions planned as part of the orthodontic treatment,
* Patients with skeletal Class I malocclusion, with an ANB angle between 0 and 4 degrees,
* Crowding in the upper and lower dental arches ranging between 1 and 6 mm,
* No missing teeth,
* No structural problems on the enamel surfaces of the teeth.

Exclusion Criteria:

* The individual has a serious systemic condition,
* The individual shows insufficient cooperation with orthodontic treatment,
* Inadequate maintenance of oral hygiene,
* Individuals undergoing orthodontic treatment with removable appliances,
* Presence of severe skeletal malocclusion,
* Structural enamel defects, such as hypomineralization, in the teeth to be evaluated.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients who received orthodontic treatment at Erciyes University Faculty of Dentistry
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
L, a, b and ΔE parameters | "through study completion, an average of 1 year".
  These scans were recorded using the intraoral scanning device 3Shape Trios (3Shape Trios 3 Plus, Copenhagen, Denmark). To provide numerical data for the color analysis (L, a, b, ΔE) performed, the recordings were transferred to the Adobe Photoshop program (Adobe Inc., San Jose, California, USA).

SECONDARY OUTCOMES:
ΔF and ΔFmax parameters | "through study completion, an average of 1 year".
  The secondary outcome was that the formation (analysed by ΔF and ΔFmax parameters; loss of fluorescence) of WSLs on the buccal surfaces of the incisor, canine and premolar teeth was assessed by the QLF-D machine and software during the pre-treatment and post-treatment examination visits. QLF images were obtained to assess enamel changes in all patients pre- (T0) and post-treatment (T1).
ΔQ and WS area parameters | "through study completion, an average of 1 year".
  The secondary outcome was the development of WSLs (analysed by ΔQ and WS area parameters; with the degree of demineralization) on the buccal surfaces of the incisor, canine and premolar teeth, which was assessed by the QLF-D machine and software during the pre-treatment and post-treatment evaluations. The images were then analysed by placing an analysis patch on the stained area, ensuring that the boundaries of the patch corresponded to sound enamel.
Gingival index | "through study completion, an average of 1 year".
  The Gingival Index (GI) is a widely used clinical measure in dental research to assess the severity and presence of gingivitis (inflammation of the gums).
Periodontal index | "through study completion, an average of 1 year".
  The Periodontal Index (PI) is a clinical tool used in dental research and practice to assess the overall health of the periodontium (the supporting structures of the teeth, including the gums, periodontal ligament, cementum, and alveolar bone).

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Faculty of Dentistry, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to national and local ethical rules, data is not shared.

REFERENCES:
- [Background] Yoon HI, Bae JW, Park JM, Chun YS, Kim MA, Kim M. A Study on Possibility of Clinical Application for Color Measurements of Shade Guides Using an Intraoral Digital Scanner. J Prosthodont. 2018 Aug;27(7):670-675. doi: 10.1111/jopr.12559. Epub 2016 Nov 7. PMID 29377326
- [Background] Atilla AO, Ozturk T, Eruz MM, Yagci A. A comparative assessment of orthodontic treatment outcomes using the quantitative light-induced fluorescence (QLF) method between direct bonding and indirect bonding techniques in adolescents: a single-centre, single-blind randomized controlled trial. Eur J Orthod. 2020 Sep 11;42(4):441-453. doi: 10.1093/ejo/cjz058. PMID 31375814